CLINICAL TRIAL: NCT00159198
Title: Genetic Linkage in Amyotrophic Lateral Sclerosis and Frontotemporal Dementia
Brief Title: Amyotrophic Lateral Sclerosis and Frontotemporal Dementia
Status: Terminated | Type: Observational
Why Stopped: Completed
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle BRINDEL, Department Clinical Research of Developpement
Other Study IDs: CRC01107; P011023; NCT00140777 (obsolete NCT alias)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2008-09

CONDITIONS: Frontotemporal Dementia; Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Frontotemporal dementia; Mutations spectrum; Linkage studies; Genetic epidemiology
MeSH Terms: conditions — Frontotemporal Dementia; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with frontotemporal dementia and amyotrophic lateral sclerosis
- 2: Relatives (first and second degree) of patients presenting an association of frontotemporal dementia with amyotrophic lateral sclerosis

SUMMARY:
Amyotrophic lateral sclerosis (ALS) with frontotemporal dementia (FTD) is a rare clinical entity, in which both disorders are variably associated in the same patient or within the family. This adult-onset disorder, which is rapidly fatal, occurs in some families with autosomal dominant (AD) transmission and age-dependant penetrance. Two studies have provided evidence for linkage of this condition to chromosomes 15 (in a single family) and 9 (in five families). However, none of these loci have been yet confirmed. Through a national network of 10 centres with specialists for FTD and/or ALS, we have identified 35 probands with ALS-FTD, including 13 with a family history consistent with AD inheritance.

Mutations in the SOD1 and tau genes, respectively responsible for autosomal dominant forms of ALS and FTD, will be excluded by direct sequencing. We will then extend the pedigree of the 13 autosomal dominant families to all consenting first, second and eventually third degree relatives, using well defined criteria for FTD and ALS. The same strategy will be applied to newly identified families during the course of the project (at least, seven families with AD inheritance expected). Linkage studies will be performed in the 20 families using markers from the two candidate regions on chromosomes 9 and 15. Then, refinement of the candidate region will be obtained by analyzing the linked families with a high density of microsatellite markers. This should lead to the refinement of the candidate regions, allowing to search for mutations in candidate genes. Genes located within the critical regions will be prioritized for their analysis by sequencing, according to their expression in the nervous system and to their function.

Once the responsible gene(s) will be identified, it will then possible to define its spectrum of mutations and to establish genotype/phenotype correlations. Alternatively, if none of the candidate regions is confirmed, a genome wide search will be performed, allowing to identify one or more loci for ALS-FTD. The same strategy would then be applied to identify the corresponding gene(s). This project should contribute for identifying the molecular basis of this devastating disorder with practical consequences for genetic counselling in ALS-FTD families, and with the perspective of elucidating the pathophysiology of this disorder.

DETAILED DESCRIPTION:
The objective of this study without direct individual benefit is to confirm the linkage with one or another region of the two identified regions (chromosomes 9 and 15) or to identify a new implicated chromosomal region, and then to reduce the linkage interval in order to identify the responsible gene(s) and characterize the mutations with the study of at least 9 families with FTD and ALS.

ELIGIBILITY:
Inclusion Criteria:

* ALS with FTD, "pure" FTD but with knowledge of relatives with ALS-FTD or "pure" ALS, "pure" ALS but with knowledge of relatives with ALS-FTD or "pure" FTD (not carriers of a mutation in the tau and SOD1 genes), relatives signing the informed consent

Exclusion Criteria:

* Minors, persons refusing to sign the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and relatives coming in outcome clinics. They are all volunteers and agree to give a blood sample and signing an informed consent explaining the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2002-09; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Brice, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, University Paris 6
Locations (15):
- France (15):
  - CHU de la Côte de Nacre, Caen
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital La Timone, Marseille
  - Hôpital Sainte-Marguerite, Marseille
  - Hôpital Guillaume et René Laënnec, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Pitié-Salpêtrière - Centre du Langage-Neuropsychologie, Paris
  - Hôpital Pitié-Salpêtrière - Fédération de Neurologie, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier, Saint-Brieuc
  - Hôpital Bellevue, Saint-Etienne
  - Hôpital Civil, Strasbourg
  - Hôpital Purpan, Toulouse

REFERENCES:
- [Result] Le Ber I, Guedj E, Gabelle A, Verpillat P, Volteau M, Thomas-Anterion C, Decousus M, Hannequin D, Vera P, Lacomblez L, Camuzat A, Didic M, Puel M, Lotterie JA, Golfier V, Bernard AM, Vercelletto M, Magne C, Sellal F, Namer I, Michel BF, Pasquier J, Salachas F, Bochet J; French research network on FTD/FTD-MND; Brice A, Habert MO, Dubois B. Demographic, neurological and behavioural characteristics and brain perfusion SPECT in frontal variant of frontotemporal dementia. Brain. 2006 Nov;129(Pt 11):3051-65. doi: 10.1093/brain/awl288. PMID 17071924
- [Result] van der Zee J, Le Ber I, Maurer-Stroh S, Engelborghs S, Gijselinck I, Camuzat A, Brouwers N, Vandenberghe R, Sleegers K, Hannequin D, Dermaut B, Schymkowitz J, Campion D, Santens P, Martin JJ, Lacomblez L, De Pooter T, Peeters K, Mattheijssens M, Vercelletto M, Van den Broeck M, Cruts M, De Deyn PP, Rousseau F, Brice A, Van Broeckhoven C. Mutations other than null mutations producing a pathogenic loss of progranulin in frontotemporal dementia. Hum Mutat. 2007 Apr;28(4):416. doi: 10.1002/humu.9484. PMID 17345602
- [Result] Le Ber I, van der Zee J, Hannequin D, Gijselinck I, Campion D, Puel M, Laquerriere A, De Pooter T, Camuzat A, Van den Broeck M, Dubois B, Sellal F, Lacomblez L, Vercelletto M, Thomas-Anterion C, Michel BF, Golfier V, Didic M, Salachas F, Duyckaerts C, Cruts M, Verpillat P, Van Broeckhoven C, Brice A; French Research Network on FTD/FTD-MND. Progranulin null mutations in both sporadic and familial frontotemporal dementia. Hum Mutat. 2007 Sep;28(9):846-55. doi: 10.1002/humu.20520. PMID 17436289
- [Result] Guedj E, Le Ber I, Lacomblez L, Dubois B, Verpillat P, Didic M, Salachas F, Vera P, Hannequin D, Lotterie JA, Puel M, Decousus M, Thomas-Anterion C, Magne C, Vercelletto M, Bernard AM, Golfier V, Pasquier J, Michel BF, Namer I, Sellal F, Bochet J, Volteau M, Brice A, Meininger V; French Research Network on FTD/FTD-MND; Habert MO. Brain spect perfusion of frontotemporal dementia associated with motor neuron disease. Neurology. 2007 Jul 31;69(5):488-90. doi: 10.1212/01.wnl.0000266638.53185.e7. No abstract available. PMID 17664410
- [Result] Le Ber I, Camuzat A, Hannequin D, Pasquier F, Guedj E, Rovelet-Lecrux A, Hahn-Barma V, van der Zee J, Clot F, Bakchine S, Puel M, Ghanim M, Lacomblez L, Mikol J, Deramecourt V, Lejeune P, de la Sayette V, Belliard S, Vercelletto M, Meyrignac C, Van Broeckhoven C, Lambert JC, Verpillat P, Campion D, Habert MO, Dubois B, Brice A; French research network on FTD/FTD-MND. Phenotype variability in progranulin mutation carriers: a clinical, neuropsychological, imaging and genetic study. Brain. 2008 Mar;131(Pt 3):732-46. doi: 10.1093/brain/awn012. Epub 2008 Feb 1. PMID 18245784
- See also: Related Info — http://www.aphp.fr